CLINICAL TRIAL: NCT03595449
Title: Patient Satisfaction in Mohs Micrographic Surgery With Supplemental Lidocaine Jelly
Brief Title: Lidocaine Jelly for Pain Control During Mohs Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shari Ochoa MD, Assistant Professor, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-011142
Record Dates: First submitted 2018-04-06; First posted 2018-07-23 (Actual); Results first posted 2021-06-22 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Pain; Satisfaction, Consumer
MeSH Terms: conditions — Pain; Consumer Behavior | interventions — Lidocaine; phenylmercury borate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine jelly (Active Comparator): This is the group that will have lidocaine jelly applied during Mohs surgery
  Interventions: Drug: Lidocaine jelly
- Surgilube (Sham Comparator): This is the group that will have surgilube (placebo) applied during Mohs surgery
  Interventions: Drug: Surgilube

INTERVENTIONS:
Drug: Lidocaine jelly — lidocaine 2% jelly applied during Mohs surgery
  Other Names: lidocaine
  Arms: Lidocaine jelly
Drug: Surgilube — surgilube (placebo) applied during Mohs surgery
  Arms: Surgilube

SUMMARY:
Does the use of lidocaine jelly during Mohs surgery on the nose decrease the total amount of lidocaine used during surgery.

Does patient satisfaction improve when lidocaine jelly is used during Mohs surgery of the nose?

DETAILED DESCRIPTION:
Hypothesis: Supplementing lidocaine/epinephrine injections with intralesional lidocaine jelly will decrease the overall quantity of lidocaine/epinephrine injectable used, and will decrease patients' self-reported pain/anxiety associated with needle sticks.

Objectives: To assess how using lidocaine jelly in Mohs surgery impacts 1) the overall quantity of lidocaine/epinephrine injectable needed to maintain anesthesia, and 2) patients' pain/anxiety associated with anesthesia injections.

Background:

Mohs micrographic surgery is a procedure that removes cancerous lesions of the skin in a step-wise fashion. Patients are injected with local analgesia for tumor extirpation. The tumor is removed and the tissue is sent for histopathology while the patient waits. Tissue processing time can take up to 2 hours during which the effects of the local analgesia have waned. Once the tissue has been process and examined, patients are brought back to the surgical suite and either have another section of tissue removed (if the margins were positive) or have the wound reconstructed (if the margins were negative). Lidocaine Hydrochloride (Xylocaine) injection with Epinephrine is the traditionally method used to maintain local anesthesia throughout the procedure. The FDA has declared a shortage of this injectable Lidocaine/Epinephrine, stressing the need for a substitute drug. Additionally, multiple needle sticks can be uncomfortable and anxiety provoking for patients. Needle sticks on hypersensitive areas such as the nose can be particularly painful. Previous research has demonstrated that a different form of anesthetic, a topical lidocaine jelly, is efficient in prolonging anesthesia in Mohs surgery (Robins, 1991). No study has published the impact of supplemental lidocaine jelly use on the overall quantity of injection needed, nor on patient pain/anxiety associated with needle sticks.

Methods:

We will conduct a prospective, randomized trial of 250 patients receiving Mohs micrographic surgery to lesions on the nose. Annually Mohs micrographic surgery is performed on approximately 900 patients with 30% of these procedures being performed on lesions on the nose. Patients receiving Mohs treatment for lesions on the nose will be randomly assigned to one of two groups: (1) those whose wounds will be dressed with lidocaine jelly (treatment group), and (2) those whose wounds will be dressed with surgical lubricant (control/placebo group).

All patients will receive a pre-treatment baseline pain/anxiety survey followed by an initial lidocaine injection. The amount of lidocaine/epinephrine injection each patient receives throughout remaining stages of surgery will be recorded, as per the current workflow. All patients will complete a second pain/anxiety survey immediately after numbing but prior to the first stage of surgery.

After the first stage of surgery, either lidocaine jelly or surgical lubricant will be applied to the wound followed by a pressure bandage as per standard practice. Dressing are removed immediately prior to the next stage of surgery. After each subsequent stage of surgery, an identical wound dressing will be placed on the operative site.

Immediately prior to each subsequent stage of surgery, we will assess patients' pain sensation, and additional lidocaine/epinephrine will be injected if needed. After the surgical site is re-anesthetized, vital signs will be recorded and the Pain/Anxiety survey administered immediately prior to the first incision of that stage.

ELIGIBILITY:
Inclusion criteria:

Patients having Mohs surgery on the nose who are able to consent to the study >18 years old

Exclusion criteria:

unable to consent for themselves known allergy to lidocaine Mohs surgery in locations other than the nose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shari A Ochoa, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine Jelly: This group had lidocaine jelly applied during Mohs surgery
  Lidocaine jelly: lidocaine 2% jelly applied during Mohs surgery
- Surgilube: This group had surgilube (placebo) applied during Mohs surgery
  Surgilube: surgilube (placebo) applied during Mohs surgery
Period: Overall Study
Arm/Group | Lidocaine Jelly | Surgilube
Started | 118 | 115
Completed | 118 | 115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Jelly | Surgilube | Total
Number analyzed (Participants) | 118 | 115 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (10.46) | 71.7 (11.38) | 72.0 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 53 | 97
  Male | 74 | 62 | 136
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 113 | 109 | 222
  Hispanic | 2 | 0 | 2
  Asian/Pacific Islander | 0 | 1 | 1
  Other | 1 | 0 | 1
  Unknown | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 118 | 115 | 233

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Patient Perception of Pain Score
Description: The mean change of total pain score of patient perception of pain. As measured by the question "Rate the pain of your nose from 0 to 10. 0 being no pain, 10 being the worst pain of your life."
Time Frame: baseline to stage 1 of Mohs surgery, approximately one hour
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lidocaine Jelly | Surgilube
Number analyzed (Participants) | 118 | 115
score on a scale | 0.5 [0.2 to 0.8] | 0.3 [0.1 to 0.6]

2. Secondary Outcome: Mean Total Amount of Intervention (Lidocaine or Surgilube) Used
Description: The mean total amount of intervention used as measured by milligrams (mg)
Time Frame: Through completion of Mohs surgery, approximately one day
Population: Data was not collected or analyzed for four subjects in each arm
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Lidocaine Jelly | Surgilube
Number analyzed (Participants) | 111 | 114
mg | 28.1 (29.0) | 24.4 (18.80)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study, approximately one day for each subject
Arm/Group | Lidocaine Jelly | Surgilube
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/115
Other Adverse Events (participants affected / at risk) | 0/118 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT03595449/Prot_SAP_000.pdf